CLINICAL TRIAL: NCT03613792
Title: Remifentanil Plus Ketamine Versus Midazolam Plus Fentanyl for Dynamic Flexible Bronchoscopy: Randomized Double-blind Clinical Trial
Brief Title: Remifentanil Plus Ketamine for Dynamic Flexible Bronchoscopy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in procedure means limited value for study question
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Satya Krishna Ramachandran, Vice Chair of Quality and Safety, Associate Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018P000023
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Bronchoscopy
Keywords: dynamic; flexible
MeSH Terms: interventions — Remifentanil; Fentanyl; Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Remifentanil and Ketamine Group (Active Comparator): Patients in Group 1 will receive remifentanil and ketamine. Remifentanil will be administered initially with a 1mcg/kg IV bolus followed by a continuous infusion, 0.1 to 0.15 mcg/kg/min IV (using ideal body weight) with titration to a maximum dose of 0.2 to 0.4 mcg/kg/min IV. Total dose of ketamine will be titrated from 10 to 40 mg, based on clinical judgment, and it will be recorded. Ketamine will be delivered using 2mL syringes, previously filled with ketamine in normal saline at a 10mg/mL concentration.
  Interventions: Drug: Remifentanil; Drug: Ketamine
- Fentanyl and Midazolam (Active Comparator): The patients in this group will receive fentanyl doses that range between 0.5 to 2 mcg/kg (25 - 50 mcg) IV bolus in combination with midazolam 1-5 mg bolus over at least 2 minutes as determined by attending anesthesiologist (not to exceed 2.5 mg / 2 min per package insert). Total dosing of fentanyl and midazolam may be titrated, based on clinical judgment, and it will be recorded. Maintenance, additional midazolam doses of 25% of total initial dose required to achieved desired sedation may be administered IV if additional sedation is considered necessary
  Interventions: Drug: Fentanyl; Drug: Midazolam

INTERVENTIONS:
Drug: Remifentanil — Opioid analgesic
  Arms: Remifentanil and Ketamine Group
Drug: Fentanyl — Opioid analgesic
  Arms: Fentanyl and Midazolam
Drug: Midazolam — Benzodiazepine
  Other Names: Versed
  Arms: Fentanyl and Midazolam
Drug: Ketamine — Analgesic
  Arms: Remifentanil and Ketamine Group

SUMMARY:
This randomized controlled pilot clinical trial will enroll patients undergoing dynamic flexible bronchoscopy will be randomized to receive one of the two anesthetic combinations described above. The study will determine if there is a difference when considering patient and physician and satisfaction when performing DFB. Also, safety and efficacy of the two pharmacological combinations (fentanyl + midazolam and remifentanil + ketamine) used will be evaluated.

ELIGIBILITY:
Inclusion criteria:

* Adult (>18 years-old)
* Undergoing planned flexible bronchoscopy with dynamic maneuvers for Excessive Central Airway Collapse assessment at Beth Israel Deaconess Medical Center.

Exclusion criteria:

* Patients with any past medical history of disease that would put them at risk of receiving one of the four proposed medications. This includes, but it's not limited to, allergies, advanced stage kidney disease, congestive heart failure and non-controlled hypertension.
* With a known/documented history of opioid abuse at any point during life.
* PO2< 60 mmHg or SO2 <85% on room air during any of the encounters with physicians between the moment of initial screening and the procedure itself.
* PaCO2 >60 mmHg
* Planned additional procedure(s) requiring general anesthesia after the dynamic bronchoscopy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction with Sedation Instrument (PSSI) | Two hours after procedure conclusion, prior to patient discharge from the hospital
  The primary outcome will be a difference in patient satisfaction with sedation, as determined by a 5-point difference in the PSSI questionnaire. The total score will be assessed by summing the responses to each question. In the scale, 0 will denote no satisfaction (worst outcome) and 100 will represent the greatest possible satisfaction (best outcome).

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for Discomfort | Two hours after procedure conclusion, prior to patient discharge from the hospital
  Difference between both groups in terms of numerical rating scale (NRS) for discomfort associated with the procedure (as reported by the patient). In the scale, 0 will denote no discomfort (best outcome) and 5 will represent the greatest possible discomfort (worse outcome).
ALDRETE score | Two hours after procedure conclusion, prior to patient discharge from the hospital
  The ALDRETE score (global assessment of post-anesthetic condition) is used to assess patients' recovery after bronchoscopy at PACU
Clinician Satisfaction with Sedation Instrument (CSSI) | Two hours after procedure conclusion, prior to patient discharge from the hospital
  The total score will be assessed by summing the responses to each question. In the scale, 0 will denote no satisfaction (worst outcome) and 100 will represent the greatest possible satisfaction (best outcome).
Severity of Cough | Two hours after procedure conclusion, prior to patient discharge from the hospital
  A scale to address severity of cough during the procedure will be used when the bronchoscope pass through the vocal cords and at the level of the proximal trachea, distal trachea and main bronchi. This scale has three categories: Mild, single coughs; Moderate, more than one episode of cough that last less than 5 seconds; and Severe, cough more than 5 seconds
Incidence of Complications | Two hours after procedure conclusion, prior to patient discharge from the hospital
  Complications such as desaturation, hypotension, pain, nausea, bradycardia, need for artificial airway or mechanical ventilation and need to abort bronchoscopy will be documented. These will then be compared as percentage of complications.
Duration of Dynamic Flexible Bronchoscopy | Two hours after procedure conclusion, prior to patient discharge from the hospital
  Defined as the total time spent between initial insertion of flexible bronchoscope and final withdrawal of such.
PACU Length of Stay | Until discharge from the PACU, on average one hour
  Total time of PACU stay with each of the pharmacological combinations, defined as the period of time between initial PACU arrival and final home or floor discharge.
Total Nebulized Lidocaine Dose | Until discharge from the PACU, on average one hour
  Total dose requirement of nebulized lidocaine, pain medication and cough suppressors at PACU discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Satya Krishna Ramachandran, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No